CLINICAL TRIAL: NCT06848517
Title: The Effectiveness of a Blended Synchronous and Asynchronous Telerehabilitation Program for Greek Adult Women With Urinary Incontinence. A Randomized Controlled Trial
Brief Title: Synchronous and Asynchronous Telerehabilitation for Women With Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Papanikolaou Dimitra-Tania, PhD(c), University of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Incontinence&Telerehab Methods
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Control Groups; Organization and Administration

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be kept confidential from the therapist who will administer the treatment groups. The therapist will be made aware of each patient's assignment on the first day of the intervention. The participants will remain unaware of the group to which they belong until the moment the intervention begins. Given the nature of the treatment, the intervention is not blinded between participants and therapists. However, the data analysis will be carried out by a 'blind' assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BSATP (Blended Synchronous and Asynchronous Telerehabilitation Programs) Group (Experimental): In the BSATP Group, participants will use synchronous telerehabilitation methods such as communications platforms (e.g. Zoom etc.) and asynchronous methods like educational videos (created by the researchers to meet the needs of this study). Through these, they will follow a PFM exercise treatment program at a convenient location of their choice such as their home. No face-to face meetings will take place between participants and the therapist while supervision (regarding the execution, frequency of the PFM exercises etc.) will occur remotely.
  Interventions: Other: BSATP Group
- FtFS (Face-to face Sessions) Group (Active Comparator): Participants will undertake their PFM exercise treatment in a healthcare setting under the continuous supervision of their therapist, drawing on the"realistic" treatment of UI, presently used in rehabilitation clinics etc.
  Interventions: Other: FtFS Group
- CG (Control Group) (Other): In the CG, participants will follow their PFM exercise treatment program without any supervision or face-to-face sessions with their therapist.
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Other: BSATP Group — Participants and the therapist will communicate once weekly synchronously (e.g. through video calls with a 30 minute duration), regarding the proper execution of the PFM exercises, providing motivation etc. Additionally, participants will be advised to watch the educational videos (10 mins duration) asynchronously twice a week. In total, participants will follow a BSATP three times a week (for 12 weeks). The PFM exercise program will include endurance training (slow velocity contractions), speed training (quick contractions) and "Knack maneuver" training (pre-contraction before the increment of the intra-abdominal pressure).The PFM exercise program will be based on three assessments conducted by the therapist throughout the study (baseline, 6 weeks and 12 weeks). As a result, the PFM exercise program will be individualized to meet their needs and progressively increases in difficulty, with the exercise position being modified every two weeks (e.g. supine, side, prone ect)
  Other Names: Blended Synchronous and Asynchronous Telerehabilitation Programs
  Arms: BSATP (Blended Synchronous and Asynchronous Telerehabilitation Programs) Group
Other: FtFS Group — Participants will attend one weekly face-to-face session with their therapist, to discuss the progress of their treatment and ensure its seamless continuation (intra-vaginal assessment, adjustments, motivation etc.). Each session will last approximately 30 minutes. Participants will also be advised to perform the PFM program twice a week on their own e.g. at home. In total, participants will follow a PFM program three times a week (for 12 weeks), once with their therapist and twice independently. The participants in the FtFS group will follow the same PFM exercise treatment program as the BSATP group, which will be an individualized program where the position will change every two weeks and include endurance training, speed training and 'Knack maneuver' training.
  Other Names: Face-to face Sessions
  Arms: FtFS (Face-to face Sessions) Group
Other: Control Group (CG) — The participants will be advised to follow a PFM exercise treatment program at home, based on an educational home leaflet (with instructions and images about PFM exercises) that they received during their first assessment session (baseline). The participants of this group will follow a PFM exercise therapy program (through the leaflet) which will last 12 weeks and they will be advised to attend it three times a week. No face-to-face meetings or supervision will occur by the therapist during the treatment period. Similarly to the other two intervention groups, the provided PFM exercise treatment program will be individualized, will include endurance training, speed training, and 'Knack maneuver' training, and the participants will be encouraged to change their exercise position on their own every two weeks.
  Other Names: PFM exercises without supervision
  Arms: CG (Control Group)

SUMMARY:
In the adult female Greek population,approximately 27% suffer from urinary incontinence (UI). Nowadays, the conservative, evidence-based and 'gold standard' therapy of UI involves pelvic floor muscles (PFM) training programs, which are effective when performed intensively (daily) and for at least three months' duration. Unfortunately, patients' adherence to PFM exercises programs is often compromised for various reasons (lack of patient interest, inability to exercise daily etc.). Therefore, the development of synchronous and asynchronous telerehabilitation programs has revolutionized UI treatment, because they offer an interactive environment which might increase patient motivation and improve patient's adherence to this demanding PFM exercise regime. Synchronous Telerehabilitation Programs (STP) have developed via communication platforms that allow users to connect with video, audio, phone, and chat applications (e.g. Zoom), where users can interact in real time with their therapist and follow their treatment through the PFM exercise program. Furthermore, Asynchronous Telerehabilitation Programs (ATP) have emerged via mobile applications, educational videos etc., where users can follow their treatment using the PFM exercise program at a more convenient time that fits into their personal schedule. Although some studies have examined either STP or ATP with or without face-to-face sessions, no study has investigated a blended approach of STP and ATP for the management of UI.

Given the above, the primary aim of this study is to evaluate the effectiveness of a blended STP and ATP, in comparison to face-to-face therapy sessions. A secondary objective is to investigate the level of patients' adherence, and the amount of supervision required, in a blended STP and ATP. Furthermore, the necessity of telerehabilitation programs (whether provided in a synchronous or asynchronous manner) in the field of pelvic floor dysfunctions specifically in UI, will be explored. Finally, the study will assess the usability of a telerehabilitation program (whether provided in a synchronous or asynchronous manner) in women with UI.

DETAILED DESCRIPTION:
The study is designed to be conducted with three groups.

1. st. In the Blended STP and ATP (BSATP) group, participants will use communication platforms and educational videos to follow their PFM exercise treatment. No face-to face meetings will take place between participants and the therapist while supervision will occur remotely.
2. nd.In the Face-to-face Sessions (FtFS) group, participants will follow their PFM exercise treatment in a healthcare setting under the continuous supervision of their therapist.
3. rd. In the Control Group (CG), participants will follow their PFM exercise treatment without any supervision or face-to-face sessions with their therapist.

Three assessments sessions will take place at baseline (0 week), half-way at 6 weeks and at the end of the treatment (after 12 weeks). A follow-up assessment will be conducted at 6 and 9 months after the baseline.

Participants will be selected voluntarily through the University Urology clinic, social networks (e.g. facebook), etc. This study has been approved by the Research Ethics Committee (R.E.C.). All participants' data will be archived anonymously in a secure cloud platform accessible only to members of the research team.

To guarantee complete allocation concealment of the groups, a randomization process will be employed by a 'blind' researcher with no knowledge of the assessment or treatment procedures. The distribution of the participants to the three groups will be undertaken through a pre-defined computer-generated list, in blocks of six people. Each participant will receive a randomly assigned number from the list (through sealed envelopes), after which participants will be randomly assigned to one of the three groups using sealed envelopes.To accomplish a homogeneous sample distribution between the groups, each block will encompass three envelopes for every group. Given the nature of the treatment, the intervention is not blinded between participants and therapists. However, the data analysis will be carried through a 'blind' assessor.

An intention-to-treat analysis will performed, based on the initial allocation of participants into groups. The data will be gathered in excel tables and through Statistical Package for the Social Sciences (SPSS) version 24.0 for Windows. An analysis within the groups before and after the intervention, will be conducted using repeated measurements ANOVA. An analysis between the groups after the intervention will be carried out by the Student t-test (independent measurements). Furthermore, the effect size with 95% confidence intervals will be measured for each outcome measure with continuous variables. Results will be deemed statistically significant if p<.05. Finally, the results will be provided by means (M) values and their standard deviations (SD).

ELIGIBILITY:
Inclusion Criteria:

* Greek women,
* 18-75 years old,
* Diagnosis of Stress Urinary Incontinence (SUI) or Mixed UI (via Urodynamic examination).
* Writing and reading of the Greek language
* Having ease in using synchronous communication platforms (e.g., Zoom) and asynchronous educational videos via smart phones, tablets, computers etc
* Able to voluntarily contract the PFM, during the initial clinical examination.

Exclusion Criteria:

* 6 months after postpartum,
* Systemic diseases
* Malignancy,
* Major gynecological surgery (i.e. total hysterectomy) over the last 10 years,
* Neurological dysfunction,
* Mental impairment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on biological gender
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form (ICIQ-UI-SF) | At baseline (0 weeks), in the middle (6 weeks), at the end of the intervention (12 weeks), and at 6 and 9 months after baseline during the follow-up period
  The ICIQ-UI-SF is a patient-centered questionnaire. It includes questions that evaluate the frequency, severity, and impact of incontinence. The ICIQ-UI SF (range 0-21) is assessed using four scoring categories: (a) slight symptoms (1-5), (b) moderate symptoms (6-12), (c) severe symptoms (13-18) and (d) very severe symptoms (19-21).
1-hour Pad test | At baseline (0 week) and at the end of the intervention (12 weeks)
  The 1-hour Pad test is a clinician-administered test. The pad is weighed, the participant wear the pad and executes a set of standardized exercises (squats, running on the spot etc.). After one hour the pad re-weighed and estimated the difference in the amount of urine leakage before and after the exercises in the pad.Τhe 1-hour Pad test is assessed using three scoring categories:(a) mild incontinence (<10 ml), (b) moderate incontinence (11-50ml) and (c) severe incontinence (>50 ml)

SECONDARY OUTCOMES:
PERFECT assessment scheme | At baseline (0 week), in the middle (6 weeks), and at the end of the intervention (12 weeks)
  The PERFECT assessment scheme is a clinician-administered test. PERFECT assessment scheme will be used for digital intravaginal evaluation of PFM contraction. It assesses a) the PFMs' Power (via Modified Oxford scale) b) the PFMs' Endurance, c) the number of Repetitions the Maximum Voluntary Contraction (MVC) is performed d) the number of fast PFM contractions the participant is able to complete) the elevation of the PFMs, f) the co-contraction with other muscles (like lower abdominals) and g) the involuntary contraction of the PFM on coughing
Electromyographic (EMG) PFM's activity | At baseline (0 week), in the middle (6 weeks), and at the end of the intervention (12 weeks)
  The EMG is a clinician-administered test. The intravaginal probe is inserted into the vagina to measure the PFMs electromyographic (EMG) activity of the PFM contraction, displaying the results on the computer as feedback (NeuroTrac® Software). Similarly to the PERFECT assessment scheme above, it evaluates the following PFM parameters: endurance, repetitions, fast contractions and involuntary PFM contraction during coughing.
Australian Pelvic Floor Questionnaire (APFQ) | At baseline (0 weeks), at the end of the intervention (12 weeks), and at 6 and 9 months after baseline during the follow-up period
  The APFQ is a patient-centered questionnaire. Australian Pelvic Floor Questionnaire (APFQ), which is standardized in the Greek language, evaluates 42 questions in four categories: bladder (1-15 question), bowel ( 16-27 question), pelvic organ prolapsed (28-32 question) and sexual function (33-42 question).The scores for each category are calculated by dividing the total score by the number of relevant questions and multiplying by 10. As a result, the scores for each area range from 0 to 10 with a total score ranging from 0 to 40 (2 questions are not included in the total score). A higher score reflects more severe symptoms
Patient Global Impression of Improvement (PGI-I Scale) | At the end of the intervention (12 weeks)
  The PGI-I Scale is a patient-centered questionnaire. The participants evaluate their perceived improvement on a scale from 1 ('much better') to 7 ('much worse').
Adherence Questionnaire (AQ) | At the middle (6 weeks), and at the end of the intervention (12 weeks)
  The AQ is a patient-centered questionnaire. It includes 28 questions in total and most of them are closed type (yes/no). It is categorized into the following sections: a) social and demographic factors (1 to 4 questions), b) therapy-related factors (5 to 9 questions) c) healthcare team and system-related factors (physical therapists) (10 to 12 questions), d) patient-related factors (13 to 23 questions) and e) condition-related factors (24 to 26 questions). Question 27 pertains to a 10-point scale of adherence while question 28 pertains to an open-ended answer where the patient explains the reason of low or moderate adherence.
Adherence Exercise Diary (AED) | At baseline (0 week) the PFM AED is supplied to the participants, who will then re-submit it at the end of the intervention(12 weeks)
  A PFM AED, designed to meet the needs of the current research. Participants record the daily and weekly frequency of performing the PFM exercises, along with the sets, repetitions and the rest periods they follow throughout their treatment.
Telehealth Usability Questionnaire (TUQ) | At the end of the intervention(12 weeks)
  The Telehealth Usability Questionnaire (TUQ) is a patient-centered questionnaire, standardized in the Greek language, and consists of 21 questions. The patients rate their opinion on a scale from 1 ('strongly disagree') to 7 ('strongly agree'). The total score is calculated and then the average of the responses to all statements, is determined. The higher the total average, the higher the usability of the telehealth system.
"The Necessity of Creating Tele-rehabilitation Services for Pelvic Floor Dysfunctions (PFD)" through a Questionnaire | At baseline (0 weeks)
  It is a patient-centered questionnaire, which was developed in the Greek language and underwent pilot testing as part of a Master's dissertation. It was created through a multi-stage process. The questionnaire consists of 23 items which are divided into the following 5 sections: a) Socio-demographic questions, b) questions regarding technology, c) questions regarding participants' intention to use telerehabilitation programs for PFD d) questions related to compliance with telerehabilitation programs and e) questions regarding the cost of telerehabilitation programs for PFD. Participants respond using closed-ended multiple choice answers. Finally, the purpose of this questionnaire is to gather information regarding the extent to which women are aware of the existence of telerehabilitation services for PFD, and whether they would be willing to participate in such a program.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitra-Tania Papanikolaou, Principal Investigator — University of Patras
Locations (1):
- University of Patras, School of Health Rehabilitation Science, Department of Physiotherapy, Pátrai, Rion, Achaia, Greece

REFERENCES:
- [Background] Papanikolaou DT, Lampropoulou S, Giannitsas K, Skoura A, Fousekis K, Billis E. Pelvic floor muscle training: Novel versus traditional remote rehabilitation methods. A systematic review and meta-analysis on their effectiveness for women with urinary incontinence. Neurourol Urodyn. 2023 Apr;42(4):856-874. doi: 10.1002/nau.25150. Epub 2023 Feb 18. PMID 36808744